CLINICAL TRIAL: NCT05285345
Title: Implementation of a Consensus-Based Discharge Protocol for Preterm Infants With Lung Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jonathan Levin, Instructor of Pediatrics, Boston Children's Hospital
Other Study IDs: IRB-P00039393
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary Dysplasia; NICU Discharge
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Guideline Implementation: Participants in this group will be recruited during the first 3 months of the study and the time will be used for baseline data collection with existing standards of care around discharge practices of infants with BPD
- Post-Guideline Implementation: After 3 months, the discharge bundle developed from consensus from the Delphi process will be introduced to both NICUs using Quality Improvement principles. Participants will be recruited after the introduction of the discharge bundle.

SUMMARY:
The researchers have worked to create consensus recommendations among national efforts to help with the transition and coordination of care for preterm infants with lung disease around discharge from the neonatal intensive care unit to home. This study looks to evaluate implementation of the recommendations at Boston Children's Hospital and referring NICU's (Beth Israel Deaconess Medical Center and Brigham and Women's Hospital). Specifically, the research team will be looking at follow-up rates, healthcare utilization, and parental satisfaction/feedback with implementation of these guidelines.

DETAILED DESCRIPTION:
Premature infants with bronchopulmonary dysplasia (BPD) have complex care needs around discharge. BPD affects up to 40% of former preterm infants born at <28 weeks gestation, with about 10,000 new cases of BPD in the United States every year. Healthcare utilization in this population in the first two years of life is high, with increased hospitalizations, visits, and medication usage. Coordinated follow-up programs may help improve outcomes and reduce rates of hospitalization in this population. However, guidelines do not exist to identify which infants discharging from the NICU should be targeted for specialty follow-up for their respiratory disease, the time frame and format that this should occur, and which evaluations should be performed routinely around discharge.

This will be an implementation study, measuring outcomes 3 months prior and 3 months after enactment of a discharge bundle for preterm infants with BPD at local NICUs (Brigham and Women's Hospital, Beth Israel Deaconess Medical Center) who will be followed by Boston Children's Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born <32 weeks with at least mild BPD, defined as 28 days of respiratory support after birth.
* Efforts will be made to include a mix of infants with mild, moderate, and severe BPD, including infants discharged on oxygen.

Exclusion Criteria:

* Discharge to a location other than home.
* Infants with other congenital disease (cardiac, genetic, neurological) thought to contribute significantly to their respiratory disease.

Ages: 0 Days to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This will be an implementation study, measuring outcomes 3 months prior and 3 months after enactment of a discharge bundle for preterm infants with BPD at local NICUs (Brigham and Women's Hospital, Beth Israel Deaconess Medical Center) who will be followed by Boston Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Healthcare Utilization | 8 months
  Review of emergency encounters, urgent care visits, and hospital readmissions in the first 6 months after NICU discharge.

SECONDARY OUTCOMES:
Rates of pulmonary follow-up and use of telemedicine in follow-up | 8 months
  Review of medical record
Completion of recommended evaluations and testing | 8 months
  Review of medical record
Medication use | 8 months
  Review of medical record
Home oxygen use | 8 months
  Review of medical record
Feeding | 8 months
  Review of medical record
Family satisfaction with care for respiratory symptoms around and after discharge | 8 months
  Assessed by surveys

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Levin, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States